CLINICAL TRIAL: NCT00929006
Title: Study to Assess Acute Progesterone Suppression of Wake vs. Sleep Luteinizing Hormone Pulse Frequency in Pubertal Girls With and Without Hyperandrogenism
Brief Title: Acute Progesterone Suppression of Wake vs. Sleep Luteinizing Hormone Pulse Frequency in Pubertal Girls With and Without Hyperandrogenism
Acronym: CRM003
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Professor of Pediatrics, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 13717
Record Dates: First submitted 2009-06-23; First posted 2009-06-26 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Puberty; Hyperandrogenism
Keywords: hyperandrogenemia; pubertal; polycystic ovary syndrome
MeSH Terms: conditions — Hyperandrogenism; Polycystic Ovary Syndrome | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Micronized progesterone suspension (Experimental): Micronized progesterone 0.8 mg/kg at 0700, 1500, 2300 and 0700 h. Progesterone is a natural hormone.
  Interventions: Drug: Micronized progesterone suspension
- Placebo (Placebo Comparator): Placebo contains only inert ingredients and is not expected to exert any direct physiological effects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Micronized progesterone suspension — Micronized progesterone 0.8 mg/kg at 0700, 1500, 2300 and 0700 h. Progesterone is a natural hormone.
  Other Names: Progesterone
  Arms: Micronized progesterone suspension
Drug: Placebo — Placebo contains only inert ingredients and is not expected to exert any direct physiological effects
  Arms: Placebo

SUMMARY:
The purpose of this study is two-fold. (1) We will determine if in mid- to late pubertal girls without hyperandrogenism (HA), progesterone (P4) acutely reduces waking luteinizing hormone (LH) frequency to a greater extent than sleep-associated LH frequency. (2) We will determine if in mid- to late pubertal girls with HA, P4 will acutely suppress waking LH frequency to a lesser degree than it does in girls without HA.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded crossover study to test the following hypotheses: (1) In normal mid- to late pubertal girls without hyperandrogenism (HA), progesterone acutely suppresses waking LH pulse frequency more than sleep-associated LH pulse frequency; and (2) compared to normal mid- to late pubertal girls without HA, acute progesterone suppression of waking LH pulse frequency is impaired in mid- to late pubertal girls with HA. Studies will be performed in mid- to late pubertal girls (at least Tanner breast stage 3 but no more than 2 years postmenarcheal). Subjects will complete two 18-hour Clinical Research Unit (CRU) admissions in separate menstrual cycles. Immediately before and during the first CRU admission, either oral micronized progesterone (0.8 mg/kg/dose) or placebo (randomized) will be given at 0700, 1500, 2300, and 0700 h. During the CRU admission, blood will be obtained every 10 minutes through an indwelling iv catheter from 1800 to 1200 h. This will allow full characterization of pulsatile LH secretion in addition to other hormone measurements. A second CRU admission (performed at least 2 months later given blood withdrawal limits) will be identical to the first except that placebo will exchanged for progesterone or vice versa (treatment crossover). The primary endpoint is LH pulse frequency while awake. (LH pulse frequency while asleep is an important secondary endpoint.) Results in pubertal girls without HA were recently published (Kim et al, J Clin Endocrinol Metab 2018;103:1112-1121). Data from girls with HA will be compared to recently-published results in girls without HA. Mean LH pulse frequency while awake will be analyzed via a hierarchical linear mixed model (HLMM). HA status (HA vs. non-HA), sleep status (wake vs. sleep), and treatment (progesterone vs. placebo) will represent fixed-effects, along with all associated interactions. Random effects will be used to account for hierarchical variance-covariance structure of the crossover study design. With regard to hypothesis testing, the association between HA status and wake LH pulse frequency will be evaluated via linear contrasts of HLMM least squares pulse frequency means. The differential impact of exogenous progesterone on wake LH pulse frequency in pubertal girls with and without HA (primary analysis) will be evaluated via the same testing method. Using published and preliminary data, we determined that, if 16 pubertal girls with HA complete both admissions, we should have at least an 80% chance of detecting a 0.2 pulse/hour differential effect of P4 on wake LH pulse frequency between the HA and the non-HA groups with a two-sided false positive rejection rate of no more than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Mid- to late pubertal adolescent girl (at least Tanner breast stage 3, but no more than 2 years postmenarcheal)
* For girls without hyperandrogenism: serum (calculated) free testosterone concentration within the Tanner stage-specific reference range and the absence of hirsutism
* For girls with hyperandrogenism: serum (calculated) free testosterone concentration greater than the Tanner stage-specific reference range and/or unequivocal evidence for hirsutism
* General good health (excepting overweight, obesity, hyperandrogenism, and adequately-treated hypothyroidism)
* Capable of and willing to provide informed assent (adolescents under age 16 years) and/or consent (adolescents over age 16 years; custodial parents or guardians of all adolescent volunteers)
* Willing to strictly avoid pregnancy with use of reliable non-hormonal methods during the study period

Exclusion Criteria:

* Inability/incapacity to provide informed consent
* Males will be excluded (hyperandrogenism is unique to females)
* Obesity resulting from a well-defined endocrinopathy or genetic syndrome
* Positive pregnancy test or current lactation
* Evidence for non-physiologic or non-PCOS causes of hyperandrogenism and/or anovulation
* Evidence of virilization (e.g., rapidly progressive hirsutism, deepening of the voice, clitoromegaly)
* Total testosterone > 150 ng/dl, which suggests the possibility of virilizing ovarian or adrenal tumor
* DHEA-S elevation > 1.5 times the upper reference range limit. Mild elevations may be seen in adolescent HA and in PCOS, and will be accepted in these groups.
* Early morning 17-hydroxyprogesterone > 200 ng/dl measured in the follicular phase, which suggests the possibility of congenital adrenal hyperplasia (if elevated during the luteal phase, the 17-hydroxyprogesterone will be repeated during the follicular phase). NOTE: If a 17-hydroxyprogesterone > 200 ng/dl is confirmed on repeat testing, an ACTH stimulated 17-hydroxyprogesterone < 1000 ng/dl will be required for study participation.
* Abnormal thyroid stimulating hormone (TSH): Note that subjects with stable and adequately treated primary hypothyroidism, reflected by normal TSH values, will not be excluded.
* Hyperprolactinemia: Mild prolactin elevations may be seen in HA/PCOS, and elevations within 20% higher than the upper limit of normal will be accepted in this group.
* History and/or physical exam findings suggestive of Cushing's syndrome, adrenal insufficiency, or acromegaly
* History and/or physical exam findings suggestive of hypogonadotropic hypogonadism (e.g., symptoms of estrogen deficiency) including functional hypothalamic amenorrhea (which may be suggested by a constellation of symptoms including restrictive eating patterns, excessive exercise, psychological stress, etc.)
* Hematocrit < 36% and hemoglobin < 12 g/dl.
* Severe thrombocytopenia (platelets < 50,000 cells/microliter) or leukopenia (total white blood count < 4,000 cells/microliter)
* Previous diagnosis of diabetes, fasting glucose > or = 126 mg/dl, or a hemoglobin A1c > or = 6.5%
* Persistent liver panel abnormalities, with two exceptions. Mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome. Also, mild transaminase elevations may be seen in obesity/HA/PCOS; therefore, elevations < 1.5 times the upper limit of normal will be accepted in such girls.
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure, asthma requiring intermittent systemic corticosteroids, etc.)
* Decreased renal function evidenced by GFR < 60 ml/min/1.73m2
* A personal history of breast, ovarian, or endometrial cancer
* History of any other cancer diagnosis and/or treatment (with the exception of basal cell or squamous cell skin carcinoma) unless they have remained clinically disease free (based on appropriate surveillance) for five years
* History of allergy to micronized progesterone.
* Body mass index (BMI)-for-age percentile < 5% (underweight)
* Due to the amount of blood being drawn, adolescent volunteers with body weight < 25 kg will be excluded.
* Restrictions on use of other drugs or treatments: No medications known to affect the reproductive system, glucose metabolism, lipid metabolism, or blood pressure can be taken in the 2 months prior to the screening visit and in the 3 months prior to the start of the study medications. Such medications include oral contraceptive pills, progestins, metformin, systemic glucocorticoids, some antipsychotic medications, and sympathomimetics/stimulants (e.g., methylphenidate).

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2008-06 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Luteinizing hormone (LH) pulse frequency | During first CRU admission and during the second CRU admission (which occurs at least 2 months after the first)
  LH pulse frequency while awake vs. while asleep pulse frequency

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Burt Solorzano, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data from this study will be deposited in the NICHD Data and Specimen Hub "DASH." We will also provide raw study data (de-identified) as supplementary materials in manuscripts (e.g., see Kim SH, et al. Progesterone-mediated inhibition of the GnRH pulse generator: differential sensitivity as a function of sleep status. J Clin Endocrinol Metab 2018; 103: 1112-1121 [PMCID in process]).

REFERENCES:
- [Derived] Kim SH, Lundgren JA, Bhabhra R, Collins JS, Patrie JT, Burt Solorzano CM, Marshall JC, McCartney CR. Progesterone-Mediated Inhibition of the GnRH Pulse Generator: Differential Sensitivity as a Function of Sleep Status. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1112-1121. doi: 10.1210/jc.2017-02299. PMID 29300925